CLINICAL TRIAL: NCT00863057
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of Duloxetine and Methadone for the Treatment of HIV-Associated Painful Peripheral Neuropathy
Brief Title: Combination Pain Therapy in HIV Neuropathy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow rate of enrollment, which compromised the ability to meet study objectives in a timely manner.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A5252; 10636 (Registry Identifier: DAIDS ES); ACTG A5252
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Results first posted 2012-04-25 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2019-02

CONDITIONS: HIV Infections; Peripheral Neuropathy
Keywords: HIV Infections; Neuropathy; Pain
MeSH Terms: conditions — HIV Infections; Peripheral Nervous System Diseases; Pain | interventions — Duloxetine Hydrochloride; Methadone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine and methadone placebo, (Period 2, Weeks 6 to 9) duloxetine placebo and methadone, (Period 3, Weeks 11 to 14) duloxetine and methadone, (Period 4, Weeks 16 to 19) duloxetine placebo and methadone placebo
  Interventions: Drug: Duloxetine; Drug: Duloxetine placebo; Drug: Methadone; Drug: Methadone placebo
- 2 (Experimental): Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine placebo and methadone, (Period 2, Weeks 6 to 9) duloxetine placebo and methadone placebo, (Period 3, Weeks 11 to 14) duloxetine and methadone placebo, (Period 4, Weeks 16 to 19) duloxetine and methadone
  Interventions: Drug: Duloxetine; Drug: Duloxetine placebo; Drug: Methadone; Drug: Methadone placebo
- 3 (Experimental): Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine and methadone, (Period 2, Weeks 6 to 9) duloxetine and methadone placebo, (Period 3, Weeks 11 to 14) duloxetine placebo and methadone placebo, (Period 4, Weeks 16 to 19) duloxetine placebo and methadone
  Interventions: Drug: Duloxetine; Drug: Duloxetine placebo; Drug: Methadone; Drug: Methadone placebo
- 4 (Experimental): Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine placebo and methadone placebo, (Period 2, Weeks 6 to 9) duloxetine and methadone, (Period 3, Weeks 11 to 14) duloxetine placebo and methadone, (Period 4, Weeks 16 to 19) duloxetine and methadone placebo
  Interventions: Drug: Duloxetine; Drug: Duloxetine placebo; Drug: Methadone; Drug: Methadone placebo

INTERVENTIONS:
Drug: Duloxetine — During each treatment period, participants will take duloxetine in the following doses. On Days 1 to 5, participants will take one 30-mg capsule orally, once daily. On Days 6 to 28, participants will take two 30-mg capsules orally, once daily. During days 29 to 31 dosage will be reduced to one capsule daily and then discontinued on Day 32.
Drug: Duloxetine placebo — During each treatment period, participants will take duloxetine placebo in the following doses. On Days 1 to 5, participants will take one 30-mg capsule orally, once daily. On Days 6 to 28, participants will take two 30-mg capsules orally, once daily. During days 29 to 31 dosage will be reduced to one capsule daily and then discontinued on Day 32.
Drug: Methadone — During each treatment period, participants will take methadone in the following doses. On Days 1 to 5, participants will take one 5-mg capsule orally, twice daily. On Days 6 to 10, participants will take one 5-mg capsule orally, three times daily. On Days 11 to 28, participants will take two 5-mg capsules orally, three times daily. On Days 29 to 31, dosage will be one 5-mg capsule orally, three times daily. On Days 32 to 34, dosage will be decreased to one 5-mg capsule, twice daily and ultimately discontinued on Day 35.
Drug: Methadone placebo — During each treatment period, participants will take methadone placebo in the following doses. On Days 1 to 5, participants will take one 5-mg capsule orally, twice daily. On Days 6 to 10, participants will take one 5-mg capsule orally, three times daily. On Days 11 to 28, participants will take two 5-mg capsules orally, three times daily. On Days 29 to 31, dosage will be one 5-mg capsule orally, three times daily. On Days 32 to 34, dosage will be decreased to one 5-mg capsule, twice daily and ultimately discontinued on Day 35.

SUMMARY:
Neuropathy results from damage to the nerves in the feet and legs. It is usually experienced as pain, tingling or numbness. In HIV-infected people, neuropathy can result from the infection itself or be a side effect of antiretroviral treatment. The purpose of this study is to determine whether two different drugs, methadone and duloxetine, reduce neuropathy-associated pain in HIV-infected people. This study will also examine whether utilization of both of these drugs is more effective than treatment with only one.

DETAILED DESCRIPTION:
Peripheral neuropathy is now recognized as the most common neurological complication of HIV disease and its treatment. Before highly active antiretroviral therapy (HAART) was introduced, the prevalence of HIV-associated distal sensory polyneuropathy (DSP) was already estimated to be 35%, mostly contained to populations with moderate to advanced immunosuppression. Now, since the advent of HAART, the prevalence of HIV-associated neuropathy has increased to 52%, possibly due to a combination of antiretroviral toxic neuropathy (ATN), decreased mortality, and accumulated medical comorbidities.

Successful treatment of neuropathic pain is inherently difficult, and treatment of HIV-associated neuropathic pain is particularly complicated. To date, evidence supporting effective therapies for neuropathic HIV-associated pain is lacking, despite several types and classes of drugs having been evaluated in clinical trials. This study will evaluate the safety and efficacy of duloxetine, methadone, and the combination of duloxetine and methadone in painful HIV-associated neuropathy. Both of these drugs are approved by the Food and Drug Administration (FDA) but for purposes unrelated to HIV-associated neuropathy, and no previous studies have utilized these two treatments for this purpose.

For this study, 120 participants with painful HIV-associated neuropathy will be recruited. The trial will last for approximately 23 weeks. Each participant will receive a total of 4 study treatments. The following treatment pairings will be given in a sequence determined by randomization:

1. duloxetine and methadone placebo
2. methadone and duloxetine placebo
3. duloxetine and methadone
4. duloxetine placebo and methadone placebo

Each treatment period will last 4 weeks and will be followed by a 1-week combined taper and washout.

People wishing to enroll in this study will have a screening visit that will last about 3 hours. During this visit, participants will have an HIV test, physical exam, neurologic exam, blood drawn, electrocardiogram (EKG), and a pregnancy test, if applicable. Participants will also be asked about their current health and any medications they may be taking. They will also be asked about their mood and be given the results of tests performed at the screening visit.

If screening qualifies participants for the study, they will return for a pre-entry visit lasting 2 hours. During this visit, participants will have a limited physical exam and be asked about changes in their health or medicines since screening. Participants will also be given a pain diary with instructions to record neuropathy pain every day for each of the 7 days before beginning the study and throughout the study.

After beginning the study, participants will return to the clinic for another 8 visits. These visits are at the end of each 4-week treatment period and at the end of each 1-week crossover period. At each visit, there will be a limited physical exam and participants will answer questions about their health and medications. Participants will also be told the results of routine lab tests and pregnancy tests performed during the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* HIV-associated neuropathy
* Able and willing to provide informed consent
* Successful completion of a daily baseline pain diary over 1 week immediately prior to entry with a mean pain intensity of 4 or more on an 11-point Likert scale
* Karnofsky performance score of 60 or more within 45 days prior to entry
* Required laboratory values. More information on this criterion can be found in the study protocol.
* Willing to comply with protocol requirements for the duration of the study, to include daily completion of the pain diary as instructed, attendance at all study visits, and avoidance of prohibited medications
* On stable or no antiretroviral therapy for 30 days prior to entry. Participants on ARV therapy should plan to remain on the same regimen and drug dose for the duration of the study. Participants not on ARV therapy should have no plans to initiate therapy during study enrollment.
* Not pregnant

Exclusion Criteria:

* Conditions that confound a diagnosis of HIV-associated neuropathy or preclude accurate assessment of neuropathy symptoms, at the discretion of the site investigator. More information on this criterion can be found in the study protocol.
* Potential for unstable neuropathy symptoms during study participation due tthe following: (1) discontinuation of dideoxynucleoside nucleoside reverse transcriptase inhibitor (NRTI) within 16 weeks prior to entry, (2)treatment within 120 days prior to entry with any drug that the site investigator considers may contribute to sensory neuropathy
* Current history of significant depression on antidepressant therapy precluding withdrawal from antidepressants, upon impression of site investigator with input from the participant's mental health provider where available
* History of active substance abuse or dependence identified through medical chart review or self-report such that, in the opinion of the site investigator, participation poses undue risk for the participant
* History of alcohol-related complications within 6 months prior to entry that include but are not restricted to alcohol withdrawal seizures, alcoholic hallucinosis, delirium tremens, or being in an alcohol detoxification program - Treatment with tricyclic antidepressants, selective serotonin reuptake inhibitors, selective norepinephrine reuptake inhibitors (SNRIs), bupropion, or tramadol that, upon judgment of the site investigator, cannot be tapered and discontinued prior to the pre-entry visit
* Treatment with an analgesic opioid regimen of more than 60 mg oral morphine equivalent per day within 45 days prior to entry
* Cognitive impairment that, in the opinion of the site investigator and based on clinical impression, might impact the ability to comply with the study protocol
* Use of an investigational agent within 45 days prior to entry except for expanded-access drugs or drugs used in an ACTG protocol for HIV treatment or for HIV-associated complications, if the drug is not prohibited by this protocol
* Acute active AIDS-defining opportunistic infection (OI) within 30 days prior to entry. Participants with no evidence of active disease and receiving maintenance therapy of AIDS-related OIs will be eligible
* Serious illness requiring systemic treatment and/or hospitalization within 45 days prior to entry
* End-stage renal dialysis requiring hemodialysis
* History of known or suspected hepatic cirrhosis diagnosed by signs and symptoms, radiography, or prior liver biopsy with Metavir score of more than 2
* Prolonged QTc interval (more than 0.45 seconds) within 90 days prior to entry
* Felt to be at high risk of opioid-induced respiratory compromise. More information on this criterion can be found in the study protocol.
* Diagnosis of a new seizure disorder or seizure within 90 days prior to entry
* History of acute angle-closure glaucoma, at the discretion of the site investigator
* Known allergy/sensitivity or any hypersensitivity to duloxetine, methadone, acetaminophen, or their ingredients
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-05 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David B. Clifford, MD, Study Chair — Washington University School of Medicine; Taylor B. Harrison, MD, Study Chair — Emory University, Department of Neurology, Neuromuscular Division
Locations (8):
- United States (8):
  - Ucsd, Avrc Crs, San Diego, California
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Northwestern University CRS, Chicago, Illinois
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - MetroHealth CRS, Cleveland, Ohio
  - Houston AIDS Research Team CRS, Houston, Texas

REFERENCES:
- [Background] Evans SR, Clifford DB, Kitch DW, Goodkin K, Schifitto G, McArthur JC, Simpson DM. Simplification of the research diagnosis of HIV-associated sensory neuropathy. HIV Clin Trials. 2008 Nov-Dec;9(6):434-9. doi: 10.1310/hct0906-434. PMID 19203909
- [Background] Valcour V, Yeh TM, Bartt R, Clifford D, Gerschenson M, Evans SR, Cohen BA, Ebenezer GJ, Hauer P, Millar L, Gould M, Tran P, Shikuma C, Souza S, McArthur JC; AIDS Clinical Trials Group (ACTG) 5157 protocol team. Acetyl-l-carnitine and nucleoside reverse transcriptase inhibitor-associated neuropathy in HIV infection. HIV Med. 2009 Feb;10(2):103-10. doi: 10.1111/j.1468-1293.2008.00658.x. PMID 19200173
- [Derived] Harrison T, Miyahara S, Lee A, Evans S, Bastow B, Simpson D, Gilron I, Dworkin R, Daar ES, Wieclaw L, Clifford DB; ACTG A5252 Team. Experience and challenges presented by a multicenter crossover study of combination analgesic therapy for the treatment of painful HIV-associated polyneuropathies. Pain Med. 2013 Jul;14(7):1039-47. doi: 10.1111/pme.12084. Epub 2013 Apr 8. PMID 23565581
- See also: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 (Clarification, August 2009) — https://rsc.tech-res.com/clinical-research-sites/safety-reporting/daids-grading-tables

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited across 8 of 15 study sites in the AIDS Clinical Trials Group system between August 2009 and October 2010. The sites were: Harbor-UCLA Medical Center, Harvard MGH, Houston AIDS Research Team, Metrohealth Medical Center in Cleveland, Northwestern University, UC San Diego Medical Center, Washington Univ., Univ. of Colorado.
Groups:
- D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P: Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine(D) and methadone placebo (MTD-P), (Period 2, Weeks 6 to 9) duloxetine placebo(D-P) and methadone(MTD), (Period 3, Weeks 11 to 14) duloxetine(D) and methadone(MTD), (Period 4, Weeks 16 to 19) duloxetine placebo(D-P) and methadone placebo(MTD-P)
  Methadone and matching placebo were initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Duloxetine and matching placebo were initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD: Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine placebo and methadone, (Period 2,Weeks6 to9)duloxetine placebo and methadone placebo, (Period 3, Weeks 11 to 14)duloxetine and methadone placebo, (Period 4, Weeks 16 to 19) duloxetine and methadone
  Methadone and matching placebo were initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6, and thereafter titrated to target dose of 10mg TID by Day 11. Duloxetine and matching placebo were initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD: Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine and methadone, (Period 2, Weeks 6 to 9) duloxetine and methadone placebo, (Period 3, Weeks 11 to 14) duloxetine placebo and methadone placebo, (Period 4, Weeks 16 to 19) duloxetine placebo and methadone
  Methadone and matching placebo were initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6, and thereafter titrated to target dose of 10mg TID by Day 11. Duloxetine and matching placebo were initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P: Participants will receive treatment in the following order: (Period 1, Weeks 1 to 4) duloxetine placebo and methadone placebo, (Period 2, Weeks 6 to 9) duloxetine and methadone, (Period 3, Weeks 11 to 14) duloxetine placebo and methadone, (Period 4, Weeks 16 to 19) duloxetine and methadone placebo
  Methadone and matching placebo were initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Duloxetine and matching placebo were initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
Period: Milestones Period 1 (Weeks 0-5)
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Started | 4 | 4 | 3 | 4
Completed | 3 | 2 | 3 | 3
Not Completed | 1 | 2 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 1 | 0 | 0
Period: Period 2 (Weeks 6-10)
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Started | 3 | 2 | 3 | 3
Completed | 3 | 1 | 2 | 2
Not Completed | 0 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Period: Period 3 (Weeks 11-15)
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Started | 3 | 1 | 2 | 2
Completed | 3 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0
Period: Period 4 (Weeks 16-20)
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Started | 3 | 1 | 2 | 2
Completed | 3 | 1 | 2 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P | Total
Number analyzed (Participants) | 4 | 4 | 3 | 4 | 15
Age, Customized [Number; unit: participants]
  20-29 | 0 | 0 | 0 | 1 | 1
  30-39 | 0 | 1 | 0 | 0 | 1
  40-49 | 0 | 0 | 1 | 1 | 2
  50-59 | 3 | 2 | 1 | 2 | 8
  >= 60 | 1 | 1 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 2
  Male | 4 | 4 | 1 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 1 | 3 | 1 | 2 | 7
  Black/African American | 2 | 1 | 1 | 1 | 5
  Hispanic/Latino | 1 | 0 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 4 | 15
Baseline CD4 Counts [Mean (Standard Deviation); unit: cells/µL] | 400 (278) | 522 (328) | 867 (162) | 249 (173) | 486 (315)
Baseline CD8 Counts [Mean (Standard Deviation); unit: cells/µL] | 970 (639) [441.50 to 1498.50] | 490 (205) [347 to 633] | 1042.33 (1110) [366 to 2324] | 794.75 (534) [399 to 1190.50] | 809.73 (618) [353 to 1333]
Baseline Log10(HIV RNA Viral Load) in copies/mL [Number; unit: participants]
  <= 1.70 | 2 | 3 | 3 | 2 | 10
  =1.71 | 0 | 0 | 0 | 1 | 1
  =2.19 | 1 | 0 | 0 | 0 | 1
  =2.34 | 1 | 0 | 0 | 0 | 1
  =4.61 | 0 | 1 | 0 | 0 | 1
  =5.90 | 0 | 0 | 0 | 1 | 1
Baseline Daily Mean Pain Intensity (MPI) Scores [Mean (Standard Deviation); unit: Scores on a scale] — Pain was measured on an 11-point Likert numerical rating scale, ranging from 0="No pain" to 10="Pain as bad as you can imagine".Participants were given diary at weeks 0, 5, 10, and 15. They started diary 7 days prior to their clinic visits at 0,4,9,14,19. Each day, recorded a number from 0 to 10. These numbers were averaged by the number of days so the total range of scores is still from 0 to 10.
  Scores on a scale | 7.8 (0.5) | 6.5 (1.3) | 6 (1) | 7.3 (2.2) | 6.9 (1.4)
Baseline Night Time Mean Pain Intensity (MPI) Scores [Mean (Standard Deviation); unit: Scores on a scale] — Pain was measured on an 11-point Likert numerical rating scale, ranging from 0="No pain" to 10="Pain as bad as you can imagine".Participants were given diary at weeks 0, 5, 10, and 15. They started diary 7 days prior to their clinic visits at 0,4,9,14,19. Each day, recorded a number from 0 to 10. These numbers were averaged by the number of days so the total range of scores is still from 0 to 10.
  Scores on a scale | 7.3 (1.0) | 6.8 (1.0) | 7.3 (1.2) | 8 (1.4) | 7.3 (1.1)
Baseline Brief Pain Inventory (BPI) Interference Scores [Mean (Standard Deviation); unit: Scores on a scale] — The BPI interference scale measured level of interference with the following seven items:
  1. General activity
  2. Mood
  3. Walking ability
  4. Normal work
  5. Relations with other people
  6. Sleep
  7. Enjoyment of life
  Interference scales range from 0='Does not interfere' to 10='Completely interferes'. The overall BPI score is the mean of seven items.
  Scores on a scale | 5.6 (1.1) | 4.1 (0.5) | 4.5 (2.8) | 6.1 (3.7) | 5.1 (2.3)
Baseline Center for Epidemiologic Studies Depression (CES-D) Scores [Mean (Standard Deviation); unit: Scores on a scale] — The CES-D is a 20-item self-report rating inventory measuring characteristic attitudes and symptoms of depression. Participants were asked to score each item:(0)Rarely,(1)Occasionally,(2)Sometimes,(3)Most of time.Some items are multiplied by -1 to change direction.
  The overall CES-D score is simply the sum of 20 items. The highest possible total CES-D score is 48, and the lowest possible score is -12. The total CES-D score is considered missing if more than 4 items are not answered.
  Scores on a scale | 13 (10) | 11 (8) | 9 (9) | 16 (22) | 12 (13)

OUTCOME MEASURES:

1. Primary Outcome: Weekly Mean Pain Score Derived From Self-reported Average Daily Pain Intensity on an 11-point Likert Scale
Description: Pain was measured on an 11-point Likert numerical rating scale, ranging from 0=''No pain" to 10=''Pain as bad as you can imagine".
  Participants were given pain diaries at weeks 0, 5, 10, and 15. They started the diary 7 days prior to their clinic visits at weeks 0, 4, 9, 14, and 19. During the 7 days, each morning, they recorded their pain level due to neuropathy by circling the number that best described their neuropathy pain on average over the past 24 hours.
Time Frame: During the fourth treatment week of each treatment period
Population: The analysis was per protocol. Since this is a cross-over trial, the number of participants analyzed do not match with the ones in the flow chart.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Duloxetine and Methadone; Duloxetine and Methadone Placebo; Duloxetine Placebo and Methadone; Duloxetine Placebo and Methadone Placebo: Methadone and matching placebo were initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6, and thereafter titrated to target dose of 10mg TID by Day 11. Duloxetine and matching placebo were initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6.
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
Scores on a scale | 5.20 (2.44) [4 to 7] | 5.91 (2.47) [4 to 8] | 6.20 (2.35) [5 to 8] | 5.70 (2.16) [4 to 8]

2. Secondary Outcome: Number of Participants With 30% or More Improvement in Mean Pain Score on an 11-point Likert Scale
Description: Pain was measured on an 11-point Likert numerical rating scale, ranging from 0=''No pain" to 10=''Pain as bad as you can imagine" at baseline and over the fourth treatment week of each treatment period.
  The % of improvement was calculated as (x-y)/x,where x was the MPI score at baseline, and y was the MPI score at the end of each treatment stage.
Time Frame: At Baseline and over the fourth treatment week of each treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
participants | 2 | 2 | 2 | 2

3. Secondary Outcome: Number of Participants With 50% or More Improvement in Mean Pain Score on an 11-point Likert Scale
Description: as for outcome 2
Time Frame: At Baseline and over the fourth treatment week of each treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
participants | 2 | 2 | 1 | 2

4. Secondary Outcome: Mean Nighttime Pain Measure on an 11-point Likert Scale
Description: Pain was measured on an 11-point Likert numerical rating scale, ranging from 0=''No pain" to 10=''Pain as bad as you can imagine".
  Participants were given pain diaries at weeks 0, 5, 10, and 15. They started the diary 7 days prior to their clinic visits at weeks 0, 4, 9, 14, and 19. During the 7 days, each morning, they recorded their pain level due to neuropathy by circling the number that best described their neuropathy pain on average during the night time.
Time Frame: Over the fourth treatment week of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
Scores on a scale | 5.20 (2.35) [4 to 6] | 5.82 (2.27) [4 to 8] | 5.90 (2.33) [5 to 7] | 6.10 (2.47) [4 to 8]

5. Secondary Outcome: Pain-related Interference Measured by the Brief Pain Inventory (BPI) Interference Items
Description: The BPI interference scale measured level of interference with the following seven items:
  1. General activity
  2. Mood
  3. Walking ability
  4. Normal work
  5. Relations with other people
  6. Sleep
  7. Enjoyment of life
  Interference scales range from 0='Does not interfere' to 10='Completely interferes'. The overall BPI score is the mean of seven item with the minimum and maximal scores of 0 and 70, respectively.
Time Frame: At the fourth week of each treatment period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
Scores on a scale | 3.14 [2.57 to 4.57] | 4.14 [2.29 to 7.14] | 3.64 [3.29 to 6.71] | 3.14 [2.57 to 5.57]

6. Secondary Outcome: Quality of Life Measured by SF-36 Healthy Survey (SF-36)
Description: The data for this outcome are not available for the analysis due to an issue with a company which provides software to calculate SF-36.
Time Frame: At the fourth treatment week of each treatment period
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Emotional Functioning as Measured by the Center for Epidemiologic Studies Depression Scale (CES-D)
Description: The CES-D is a 20-item self-report rating inventory measuring characteristic attitudes and symptoms of depression. Participants were asked to score each item: (0) Rarely, (1) Occasionally, (2) Sometimes, and (3) Most of time. Some items are multiplied by -1 to change direction. The overall CES-D score is simply the sum of 20 items. The highest possible total CES-D score is 48, and the lowest possible score is -12. The total CES-D score is considered missing if more than 4 items are not answered.
Time Frame: At the fourth treatment week of each treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
Scores on a scale | 13.8 (10.9) | 13.8 (14.5) | 13.3 (10.8) | 13.3 (13.2)

8. Secondary Outcome: Patient and Clinician Global Impression of Change (PGIC and CGIC) on a 7-point Likert Scale
Description: The GIC scale is a validated instrument that consists of seven verbal descriptors on a 7-point scale:
  1. Very much improved
  2. Much improved
  3. Minimally improved
  4. No change
  5. Minimally worse
  6. Much worse
  7. Very much worse
  Participants were carefully instructed to consider the impact of study treatments on their level of neuropathic pain intensity during the baseline phase of the study.
Time Frame: At the fourth treatment week of each treatment period
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
participants
  PGIC - Very much improved | 1 | 0 | 1 | 1
  PGIC - Much improved | 4 | 1 | 2 | 1
  PGIC - Minimally improved | 2 | 4 | 4 | 4
  PGIC - No change | 3 | 6 | 2 | 4
  PGIC - Much worse | 0 | 0 | 1 | 0
  CGIC - Very much improved | 1 | 1 | 1 | 1
  CGIC - Much improved | 4 | 1 | 3 | 1
  CGIC - Minimally improved | 1 | 1 | 3 | 3
  CGIC - No change | 4 | 8 | 3 | 4
  CGIC - Much worse | 0 | 0 | 0 | 1

9. Secondary Outcome: Use of Rescue Medication (Acetaminophen)
Time Frame: During each treatment period and the subsequent cross-over (or final study week) period
Population: The analysis was per protocol. Because of a cross-over trial, the # of participants analyzed do not match with the flow chart. Any participant who took the rescue med during the study period (incl. cross-over period) was counted in this analysis. If a participant took the rescue med twice within the same period, the number is counted as one.
Measure: Number; unit: participants
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
participants
  Treatment period (1-4, 6-9, 11-14, 16-19 weeks) | 0 | 0 | 0 | 2
  Cross-over period (5, 10, 15, 20 weeks) | 1 | 0 | 1 | 1

10. Secondary Outcome: Maximum Tolerated Dose of Duloxetine and Methadone
Time Frame: During each treatment period
Population: The number below is the highest tolerated daily dose in mg based on n=12 for Methadone and n=10 for Duloxetine.
Measure: Number; unit: mg
Groups:
- Methadone: Maximum tolerated daily dose of Methadone was reported.
- Duloxetine: Maximum tolerated daily dose of Duloxetine was reported.
Arm/Group | Methadone | Duloxetine
Number analyzed (Participants) | 12 | 10
mg | 30 | 60

11. Secondary Outcome: Number of Participants With Treatment-emergent Grade 2 to 4 Adverse Events
Description: The DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004 was used (see the link to the grading table in Protocol Section)
Time Frame: From study entry to end of study at week 20 or premature study discontinuation
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
Number analyzed (Participants) | 10 | 11 | 10 | 10
Participants | 5 | 4 | 6 | 5

12. Other Pre Specified Outcome: Sensory and Affective Qualities of Pain Measured by the McGill Pain Questionnaire - Short Form (MPQ-SF)
Description: This was one of the exploratory objectives and was not analyzed as the study was terminated. We do not have any plan to analyze this endpoint in the future.
Time Frame: At the fourth treatment week of each treatment period
Population: This was one of the exploratory objectives and was not analyzed as the study was terminated.
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Methadone Trough Level and Weekly Mean Pain Scores
Description: This was one of the exploratory objectives and was not analyzed as the study was terminated. We do not have any plan to analyze this endpoint.
Time Frame: During the fourth week of each treatment period
Population: This was one of the exploratory objectives and was not analyzed as the study was terminated.
Arm/Group | D + MTD-P, Then D-P + MTD, Then D+MTD, Then D-P + MTD-P | D-P + MTD, Then D-P + MTD-P, Then D + MTD-P, Then D + MTD | D + MTD, Then D + MTD-P, Then D-P + MTD-P, Then D-P + MTD | D-P + MTD-P, Then D + MTD, Then D-P + MTD, Then D + MTD-P
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Through out the study period. Participants were followed for the duration of study period, which is 20 weeks.
Groups:
- Duloxetine and Methadone: Duloxetine was initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Methadone was initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- Duloxetine and Methadone Placebo: Duloxetine was initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Methadone placebo was initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- Duloxetine Placebo and Methadone: Duloxetine placebo was initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Methadone was initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
- Duloxetine Placebo and Methadone Placebo: Duloxetine placebo was initiated at 30mg daily for 5 days and thereafter titrated to a target dose of 60mg daily at Day 6. Methadone placebo was initiated at 5mg twice daily (BID), titrated to 5mg three times daily (TID) on Day 6,and thereafter titrated to target dose of 10mg TID by Day 11. Each treatment period lasted four weeks and was followed by a 1-week combined taper and washout. Flexible dosing allowed participants to receive either the target ceiling dose or the maximum tolerated dose of study treatments.
Arm/Group | Duloxetine and Methadone | Duloxetine and Methadone Placebo | Duloxetine Placebo and Methadone | Duloxetine Placebo and Methadone Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 4/11 | 6/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Duloxetine and Methadone (N=10) | Duloxetine and Methadone Placebo (N=11) | Duloxetine Placebo and Methadone (N=10) | Duloxetine Placebo and Methadone Placebo (N=10)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2/8 (2) | 0 (0) | 1 (1) | 0 (0)
Dreams, Abnormal (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Total Bilirubin (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sgot (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognition, Abnormal (Nervous system disorders) | 0 (0) | 0/1 (0) | 1 (1) | 0 (0)
Mental Status Change, Psychiatric (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cramp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alkaline Phosphatase (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear Abnormality (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The results should be interpreted with caution since the total sample size was much lower than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.